CLINICAL TRIAL: NCT05965609
Title: Piloting an Adaption of Cognitive Behavioral Therapy for Insomnia for Shift Workers (CBTI-Shift)
Brief Title: Optimizing Sleep Health in Nurses
Acronym: OSHIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: American Academy of Sleep Medicine (Other); Monash University (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Jessee Dietch, Principal Investigator, Oregon State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-2021-1200
Record Dates: First submitted 2023-07-12; First posted 2023-07-28 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Circadian Rhythm Sleep-Wake Disorders, Shift Work Type; Sleep Initiation and Maintenance Disorders
Keywords: insomnia; shift work; circadian rhythm; sleep psychology; behavioral sleep medicine
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants are asked to refrain from mentioning any information about the treatment they receive when interacting with the investigator or outcomes assessors. Participants are asked not to share details of their treatment with other individuals at their workplace.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBTI (Other): Cognitive Behavioral Therapy for Insomnia
  Interventions: Behavioral: CBTI
- MRTI (Other): Multicomponent Relaxation Therapy for Insomnia
  Interventions: Behavioral: MRTI

INTERVENTIONS:
Behavioral: CBTI — Intervention includes education about sleep and behavioral and cognitive strategies to improve sleep
  Other Names: Cognitive Behavioral Therapy for Insomnia
  Arms: CBTI
Behavioral: MRTI — Intervention includes education about sleep and behavioral and relaxation strategies to improve sleep
  Other Names: Multicomponent Relaxation Therapy for Insomnia
  Arms: MRTI

SUMMARY:
The aim of the proposed study is to pilot test two behavioral sleep intervention strategies for improving insomnia among night shift working nurses.

DETAILED DESCRIPTION:
Night shift nurses with insomnia who meet all study criteria will receive one of two insomnia therapies. The specific therapy for insomnia will be determine by chance (like a flip of a coin), with an equal chance to receive either cognitive-behavioral therapy for insomnia or multicomponent relaxation therapy for insomnia, both modified for shift workers. Both therapies will be conducted over telehealth by interventionists trained in behavioral sleep medicine.

ELIGIBILITY:
Inclusion Criteria:

* Current shift working nursing staff in Oregon
* Expect to continue on shift work schedule during the study
* Meets criteria for an insomnia disorder
* Elevated insomnia symptoms
* Have daily access to internet on a smartphone, tablet, or computer; and
* Can read and write in English

Exclusion Criteria:

* People with uncontrolled medical conditions
* Presence of safety risk or condition in which study participation may be ineffective or result in increased risk to safety
* Some current treatments for insomnia
* Permanent day, evening, or rotating shift schedule
* History of seizures or manic episode; or
* Current/expected pregnancy during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index | At baseline and at the post-treatment assessment (occurring at approximately 10 weeks)
  Validated questionnaire; total score range between 0 and 28, with higher numbers representing greater insomnia severity
Retention Rate | At the post-treatment assessment (occurring at approximately 10 weeks)
  Defined as [number of participants who complete minimal therapeutic dose (at least 4 sessions)] / [number of randomized participants in treatment arm]
Session Attendance | At the post-treatment assessment (occurring at approximately 10 weeks)
  For enrolled participants, attendance rates will be calculated as [number of visits attended] / [number of total visits]
Implementation Assessment Measure | At the post-treatment assessment (occurring at approximately 10 weeks)
  Validated questionnaire; total score range between 12 and 60, with higher numbers representing greater feasibility, acceptability, and appropriateness.

SECONDARY OUTCOMES:
Change in Fatigue Severity Scale | At baseline and at the post-treatment assessment (occurring at approximately 10 weeks)
  Validated questionnaire; total score range between 9 and 63, with higher numbers representing greater fatigue.
Change in PROMIS Sleep Related Impairment 8 item | At baseline and at the post-treatment assessment (occurring at approximately 10 weeks)
  Validated questionnaire; total score range between 8-40, with higher numbers indicating greater sleep-related wake time impairment

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Dietch, PhD, Principal Investigator — Oregon State University
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be uploaded to a data repository to make it accessible for publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available within 2 years after the publication of the results pertaining to the primary aims and will be available for at least 2 years.
Access Criteria: Data will be shared only with investigators who have a clear and rigorous analytic plan and who sign a data use agreement with the principal investigator.

REFERENCES:
- [Background] McMenamin TM. A time to work: recent trends in shift work and flexible schedules. Monthly Lab Rev. 2007;130:3.
- [Background] Torquati L, Mielke GI, Brown WJ, Kolbe-Alexander T. Shift work and the risk of cardiovascular disease. A systematic review and meta-analysis including dose-response relationship. Scand J Work Environ Health. 2018 May 1;44(3):229-238. doi: 10.5271/sjweh.3700. Epub 2017 Dec 16. PMID 29247501
- [Background] Frost P, Kolstad HA, Bonde JP. Shift work and the risk of ischemic heart disease - a systematic review of the epidemiologic evidence. Scand J Work Environ Health. 2009 May;35(3):163-79. doi: 10.5271/sjweh.1319. Epub 2009 Apr 22. PMID 19387517
- [Background] Brown DL, Feskanich D, Sanchez BN, Rexrode KM, Schernhammer ES, Lisabeth LD. Rotating night shift work and the risk of ischemic stroke. Am J Epidemiol. 2009 Jun 1;169(11):1370-7. doi: 10.1093/aje/kwp056. Epub 2009 Apr 8. PMID 19357324
- [Background] Hansen J, Lassen CF. Nested case-control study of night shift work and breast cancer risk among women in the Danish military. Occup Environ Med. 2012 Aug;69(8):551-6. doi: 10.1136/oemed-2011-100240. Epub 2012 May 29. PMID 22645325
- [Background] Jia Y, Lu Y, Wu K, Lin Q, Shen W, Zhu M, Huang S, Chen J. Does night work increase the risk of breast cancer? A systematic review and meta-analysis of epidemiological studies. Cancer Epidemiol. 2013 Jun;37(3):197-206. doi: 10.1016/j.canep.2013.01.005. Epub 2013 Feb 9. PMID 23403128
- [Background] Rao D, Yu H, Bai Y, Zheng X, Xie L. Does night-shift work increase the risk of prostate cancer? a systematic review and meta-analysis. Onco Targets Ther. 2015 Oct 5;8:2817-26. doi: 10.2147/OTT.S89769. eCollection 2015. PMID 26491356
- [Background] Lin X, Chen W, Wei F, Ying M, Wei W, Xie X. Night-shift work increases morbidity of breast cancer and all-cause mortality: a meta-analysis of 16 prospective cohort studies. Sleep Med. 2015 Nov;16(11):1381-1387. doi: 10.1016/j.sleep.2015.02.543. Epub 2015 May 11. PMID 26498240
- [Background] Karlsson B, Knutsson A, Lindahl B. Is there an association between shift work and having a metabolic syndrome? Results from a population based study of 27,485 people. Occup Environ Med. 2001 Nov;58(11):747-52. doi: 10.1136/oem.58.11.747. PMID 11600731
- [Background] Gan Y, Yang C, Tong X, Sun H, Cong Y, Yin X, Li L, Cao S, Dong X, Gong Y, Shi O, Deng J, Bi H, Lu Z. Shift work and diabetes mellitus: a meta-analysis of observational studies. Occup Environ Med. 2015 Jan;72(1):72-8. doi: 10.1136/oemed-2014-102150. Epub 2014 Jul 16. PMID 25030030
- [Background] Barger LK, Lockley SW, Rajaratnam SM, Landrigan CP. Neurobehavioral, health, and safety consequences associated with shift work in safety-sensitive professions. Curr Neurol Neurosci Rep. 2009 Mar;9(2):155-64. doi: 10.1007/s11910-009-0024-7. PMID 19268039
- [Background] Johnson AL, Jung L, Song Y, Brown KC, Weaver MT, Richards KC. Sleep deprivation and error in nurses who work the night shift. J Nurs Adm. 2014 Jan;44(1):17-22. doi: 10.1097/NNA.0000000000000016. PMID 24316614
- [Background] Lee A, Myung SK, Cho JJ, Jung YJ, Yoon JL, Kim MY. Night Shift Work and Risk of Depression: Meta-analysis of Observational Studies. J Korean Med Sci. 2017 Jul;32(7):1091-1096. doi: 10.3346/jkms.2017.32.7.1091. PMID 28581264
- [Background] Angerer P, Schmook R, Elfantel I, Li J. Night Work and the Risk of Depression. Dtsch Arztebl Int. 2017 Jul 16;114(24):404-411. doi: 10.3238/arztebl.2017.0404. PMID 28669378
- [Background] Gu F, Han J, Laden F, Pan A, Caporaso NE, Stampfer MJ, Kawachi I, Rexrode KM, Willett WC, Hankinson SE, Speizer FE, Schernhammer ES. Total and cause-specific mortality of U.S. nurses working rotating night shifts. Am J Prev Med. 2015 Mar;48(3):241-52. doi: 10.1016/j.amepre.2014.10.018. Epub 2015 Jan 6. PMID 25576495
- [Background] Bureau of Labor Statistics. Standard occupational classification groups. 2018. Retrieved from bls.gov/soc/
- [Background] Lee KA. Self-reported sleep disturbances in employed women. Sleep. 1992 Dec;15(6):493-8. doi: 10.1093/sleep/15.6.493. PMID 1475563
- [Background] Oyane NM, Pallesen S, Moen BE, Akerstedt T, Bjorvatn B. Associations between night work and anxiety, depression, insomnia, sleepiness and fatigue in a sample of Norwegian nurses. PLoS One. 2013 Aug 7;8(8):e70228. doi: 10.1371/journal.pone.0070228. eCollection 2013. PMID 23950914
- [Background] Lajoie P, Aronson KJ, Day A, Tranmer J. A cross-sectional study of shift work, sleep quality and cardiometabolic risk in female hospital employees. BMJ Open. 2015 Mar 10;5(3):e007327. doi: 10.1136/bmjopen-2014-007327. PMID 25757950
- [Background] Karhula K, Hakola T, Koskinen A, Ojajarvi A, Kivimaki M, Harma M. Permanent night workers sleep and psychosocial factors in hospital work. A comparison to day and shift work. Chronobiol Int. 2018 Jun;35(6):785-794. doi: 10.1080/07420528.2018.1466792. Epub 2018 May 15. PMID 29764221
- [Background] Givens ML, Malecki KC, Peppard PE, Palta M, Said A, Engelman CD, Walsh MC, Nieto FJ. Shiftwork, Sleep Habits, and Metabolic Disparities: Results from the Survey of the Health of Wisconsin. Sleep Health. 2015 Jun;1(2):115-120. doi: 10.1016/j.sleh.2015.04.014. PMID 26894229
- [Background] Harma M, Tenkanen L, Sjoblom T, Alikoski T, Heinsalmi P. Combined effects of shift work and life-style on the prevalence of insomnia, sleep deprivation and daytime sleepiness. Scand J Work Environ Health. 1998 Aug;24(4):300-7. doi: 10.5271/sjweh.324. PMID 9754862
- [Background] Drake CL, Roehrs T, Richardson G, Walsh JK, Roth T. Shift work sleep disorder: prevalence and consequences beyond that of symptomatic day workers. Sleep. 2004 Dec 15;27(8):1453-62. doi: 10.1093/sleep/27.8.1453. PMID 15683134
- [Background] Stepanski EJ, Perlis ML. Behavioral sleep medicine. An emerging subspecialty in health psychology and sleep medicine. J Psychosom Res. 2000 Nov;49(5):343-7. doi: 10.1016/s0022-3999(00)00171-9. PMID 11164058
- [Background] Okajima I, Komada Y, Inoue Y. A meta-analysis on the treatment effectiveness of cognitive behavioral therapy for primary insomnia. Sleep Biol Rhythms. 2011;9(1):24-34.
- [Background] Murtagh DR, Greenwood KM. Identifying effective psychological treatments for insomnia: a meta-analysis. J Consult Clin Psychol. 1995 Feb;63(1):79-89. doi: 10.1037//0022-006x.63.1.79. PMID 7896994
- [Background] Morin CM, Culbert JP, Schwartz SM. Nonpharmacological interventions for insomnia: a meta-analysis of treatment efficacy. Am J Psychiatry. 1994 Aug;151(8):1172-80. doi: 10.1176/ajp.151.8.1172. PMID 8037252
- [Background] Geiger-Brown JM, Rogers VE, Liu W, Ludeman EM, Downton KD, Diaz-Abad M. Cognitive behavioral therapy in persons with comorbid insomnia: A meta-analysis. Sleep Med Rev. 2015 Oct;23:54-67. doi: 10.1016/j.smrv.2014.11.007. Epub 2014 Nov 29. PMID 25645130
- [Background] Taylor DJ, Pruiksma KE. Cognitive and behavioural therapy for insomnia (CBT-I) in psychiatric populations: a systematic review. Int Rev Psychiatry. 2014 Apr;26(2):205-13. doi: 10.3109/09540261.2014.902808. PMID 24892895
- [Background] Smith MT, Huang MI, Manber R. Cognitive behavior therapy for chronic insomnia occurring within the context of medical and psychiatric disorders. Clin Psychol Rev. 2005 Jul;25(5):559-92. doi: 10.1016/j.cpr.2005.04.004. PMID 15970367
- [Background] Dietch J, Wu J, Slavish D, et al. Characteristics of participants in trials of cognitive-behavioral therapy for insomnia: a systematic review and data synthesis. Pre-registered at PROSPERO (ID: CRD42020159476). In preparation.
- [Background] Jarnefelt H, Lagerstedt R, Kajaste S, Sallinen M, Savolainen A, Hublin C. Cognitive behavioral therapy for shift workers with chronic insomnia. Sleep Med. 2012 Dec;13(10):1238-46. doi: 10.1016/j.sleep.2012.10.003. Epub 2012 Nov 16. PMID 23168269
- [Background] Jarnefelt H, Harma M, Sallinen M, Virkkala J, Paajanen T, Martimo KP, Hublin C. Cognitive behavioural therapy interventions for insomnia among shift workers: RCT in an occupational health setting. Int Arch Occup Environ Health. 2020 Jul;93(5):535-550. doi: 10.1007/s00420-019-01504-6. Epub 2019 Dec 18. PMID 31853633
- [Background] Peter L, Reindl R, Zauter S, Hillemacher T, Richter K. Effectiveness of an Online CBT-I Intervention and a Face-to-Face Treatment for Shift Work Sleep Disorder: A Comparison of Sleep Diary Data. Int J Environ Res Public Health. 2019 Aug 24;16(17):3081. doi: 10.3390/ijerph16173081. PMID 31450619
- [Background] Vallières A, Roy M, Bastille-Denis E, Claveau S, Simon T. Exploring a behavioural therapy for insomnia in shift workers. J Sleep Disord Ther. 2015;4(202);2167-0277.
- [Background] Koffel EA, Koffel JB, Gehrman PR. A meta-analysis of group cognitive behavioral therapy for insomnia. Sleep Med Rev. 2015 Feb;19:6-16. doi: 10.1016/j.smrv.2014.05.001. Epub 2014 May 14. PMID 24931811
- [Background] Battle DE. Diagnostic and Statistical Manual of Mental Disorders (DSM). Codas. 2013;25(2):191-2. doi: 10.1590/s2317-17822013000200017. No abstract available. PMID 24413388
- [Background] Morgenthaler TI, Lee-Chiong T, Alessi C, Friedman L, Aurora RN, Boehlecke B, Brown T, Chesson AL Jr, Kapur V, Maganti R, Owens J, Pancer J, Swick TJ, Zak R; Standards of Practice Committee of the American Academy of Sleep Medicine. Practice parameters for the clinical evaluation and treatment of circadian rhythm sleep disorders. An American Academy of Sleep Medicine report. Sleep. 2007 Nov;30(11):1445-59. doi: 10.1093/sleep/30.11.1445. PMID 18041479
- [Background] Arendt J. Shift work: coping with the biological clock. Occup Med (Lond). 2010 Jan;60(1):10-20. doi: 10.1093/occmed/kqp162. PMID 20051441
- [Background] Spielman AJ, Saskin P, Thorpy MJ. Treatment of chronic insomnia by restriction of time in bed. Sleep. 1987 Feb;10(1):45-56. PMID 3563247
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Bei B, Wiley JF, Trinder J, Manber R. Beyond the mean: A systematic review on the correlates of daily intraindividual variability of sleep/wake patterns. Sleep Med Rev. 2016 Aug;28:108-24. doi: 10.1016/j.smrv.2015.06.003. Epub 2015 Jul 2. PMID 26588182
- [Background] Ganesan S, Magee M, Stone JE, Mulhall MD, Collins A, Howard ME, Lockley SW, Rajaratnam SMW, Sletten TL. The Impact of Shift Work on Sleep, Alertness and Performance in Healthcare Workers. Sci Rep. 2019 Mar 15;9(1):4635. doi: 10.1038/s41598-019-40914-x. PMID 30874565
- [Background] Taylor DJ, Wilkerson AK, Pruiksma KE, Dietch JR, Wardle-Pinkston S. Structured Clinical interview for Sleep Disorders-Revised (SCISD-R). 2019. Retrieved from insomnia.arizona.edu/scisd
- [Background] Taylor DJ, Wilkerson AK, Pruiksma KE, Williams JM, Ruggero CJ, Hale W, Mintz J, Organek KM, Nicholson KL, Litz BT, Young-McCaughan S, Dondanville KA, Borah EV, Brundige A, Peterson AL; STRONG STAR Consortium. Reliability of the Structured Clinical Interview for DSM-5 Sleep Disorders Module. J Clin Sleep Med. 2018 Mar 15;14(3):459-464. doi: 10.5664/jcsm.7000. PMID 29458705
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Background] Manber R, Carney CE. Treatment plans and interventions for insomnia: a case formulation approach. Guilford Publications; 2015.
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Background] Carney CE, Edinger JD, Kuchibhatla M, Lachowski AM, Bogouslavsky O, Krystal AD, Shapiro CM. Cognitive Behavioral Insomnia Therapy for Those With Insomnia and Depression: A Randomized Controlled Clinical Trial. Sleep. 2017 Apr 1;40(4):zsx019. doi: 10.1093/sleep/zsx019. PMID 28199710
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Chung F, Abdullah HR, Liao P. STOP-Bang Questionnaire: A Practical Approach to Screen for Obstructive Sleep Apnea. Chest. 2016 Mar;149(3):631-8. doi: 10.1378/chest.15-0903. Epub 2016 Jan 12. PMID 26378880
- [Background] Manber R, Bernert RA, Suh S, Nowakowski S, Siebern AT, Ong JC. CBT for insomnia in patients with high and low depressive symptom severity: adherence and clinical outcomes. J Clin Sleep Med. 2011 Dec 15;7(6):645-52. doi: 10.5664/jcsm.1472. PMID 22171204
- [Background] Seligman ME. The effectiveness of psychotherapy. The Consumer Reports study. Am Psychol. 1995 Dec;50(12):965-74. doi: 10.1037//0003-066x.50.12.965. PMID 8561380
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] Moore CG, Carter RE, Nietert PJ, Stewart PW. Recommendations for planning pilot studies in clinical and translational research. Clin Transl Sci. 2011 Oct;4(5):332-7. doi: 10.1111/j.1752-8062.2011.00347.x. PMID 22029804
- [Background] Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res. 2011 May;45(5):626-9. doi: 10.1016/j.jpsychires.2010.10.008. Epub 2010 Oct 28. PMID 21035130
- [Background] Carter PA, Dyer KA, Mikan SQ. Sleep disturbance, chronic stress, and depression in hospice nurses: testing the feasibility of an intervention. Oncol Nurs Forum. 2013 Sep;40(5):E368-73. doi: 10.1188/13.ONF.E368-E373. PMID 23989029
- [Background] Fiorentino L, McQuaid JR, Liu L, Natarajan L, He F, Cornejo M, Lawton S, Parker BA, Sadler GR, Ancoli-Israel S. Individual cognitive behavioral therapy for insomnia in breast cancer survivors: a randomized controlled crossover pilot study. Nat Sci Sleep. 2010 Dec 16;2:1-8. doi: 10.2147/nss.s8004. Print 2010. PMID 23616695
- [Background] Pruiksma KE, Taylor DJ, Mintz J, Nicholson KL, Rodgers M, Young-McCaughan S, Hall-Clark BN, Fina BA, Dondanville KA, Cobos B, Wardle-Pinkston S, Litz BT, Roache JD, Peterson AL; STRONG STAR Consortium. A pilot randomized controlled trial of cognitive behavioral treatment for trauma-related nightmares in active duty military personnel. J Clin Sleep Med. 2020 Jan 15;16(1):29-40. doi: 10.5664/jcsm.8116. Epub 2019 Nov 26. PMID 31957648
- [Background] Taylor DJ, Zimmerman MR, Gardner CE, Williams JM, Grieser EA, Tatum JI, Bramoweth AD, Francetich JM, Ruggero C. A pilot randomized controlled trial of the effects of cognitive-behavioral therapy for insomnia on sleep and daytime functioning in college students. Behav Ther. 2014 May;45(3):376-89. doi: 10.1016/j.beth.2013.12.010. Epub 2014 Jan 3. PMID 24680232
- [Background] Harvey AG, Soehner AM, Kaplan KA, Hein K, Lee J, Kanady J, Li D, Rabe-Hesketh S, Ketter TA, Neylan TC, Buysse DJ. Treating insomnia improves mood state, sleep, and functioning in bipolar disorder: a pilot randomized controlled trial. J Consult Clin Psychol. 2015 Jun;83(3):564-77. doi: 10.1037/a0038655. Epub 2015 Jan 26. PMID 25622197
- [Background] Tang NK, Goodchild CE, Salkovskis PM. Hybrid cognitive-behaviour therapy for individuals with insomnia and chronic pain: a pilot randomised controlled trial. Behav Res Ther. 2012 Dec;50(12):814-21. doi: 10.1016/j.brat.2012.08.006. Epub 2012 Sep 10. PMID 23123531
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- [Background] Bureau of Labor Statistics UDoL. Occupational Outlook Handbook, Registered Nurses. 2020.
- [Background] Horowitz TS, Cade BE, Wolfe JM, Czeisler CA. Efficacy of bright light and sleep/darkness scheduling in alleviating circadian maladaptation to night work. Am J Physiol Endocrinol Metab. 2001 Aug;281(2):E384-91. doi: 10.1152/ajpendo.2001.281.2.E384. PMID 11440916
- [Background] Boivin DB, James FO. Circadian adaptation to night-shift work by judicious light and darkness exposure. J Biol Rhythms. 2002 Dec;17(6):556-67. doi: 10.1177/0748730402238238. PMID 12465889
- [Background] Smith MR, Fogg LF, Eastman CI. A compromise circadian phase position for permanent night work improves mood, fatigue, and performance. Sleep. 2009 Nov;32(11):1481-9. doi: 10.1093/sleep/32.11.1481. PMID 19928387
- [Background] Minors DS, Waterhouse JM. Does 'anchor sleep' entrain circadian rhythms? Evidence from constant routine studies. J Physiol. 1983 Dec;345:451-67. doi: 10.1113/jphysiol.1983.sp014988. PMID 6663508
- [Background] Jackson ML, Banks S, Belenky G. Investigation of the effectiveness of a split sleep schedule in sustaining sleep and maintaining performance. Chronobiol Int. 2014 Dec;31(10):1218-30. doi: 10.3109/07420528.2014.957305. Epub 2014 Sep 15. PMID 25222346
- [Background] Vallières A, Bastille-Denis E, Morin C, Espie C. Circadian rhythm disorders II-shift work. The Oxford Handbook of Sleep and Sleep Disorders. 2012;1:626-643.
- [Background] Zee PC, Goldstein CA. Treatment of shift work disorder and jet lag. Curr Treat Options Neurol. 2010 Sep;12(5):396-411. doi: 10.1007/s11940-010-0090-9. PMID 20842597
- [Background] Huang LB, Tsai MC, Chen CY, Hsu SC. The effectiveness of light/dark exposure to treat insomnia in female nurses undertaking shift work during the evening/night shift. J Clin Sleep Med. 2013 Jul 15;9(7):641-6. doi: 10.5664/jcsm.2824. PMID 23853555
- [Background] Crowley SJ, Lee C, Tseng CY, Fogg LF, Eastman CI. Combinations of bright light, scheduled dark, sunglasses, and melatonin to facilitate circadian entrainment to night shift work. J Biol Rhythms. 2003 Dec;18(6):513-23. doi: 10.1177/0748730403258422. PMID 14667152
- [Background] Crowley SJ, Lee C, Tseng CY, Fogg LF, Eastman CI. Complete or partial circadian re-entrainment improves performance, alertness, and mood during night-shift work. Sleep. 2004 Sep 15;27(6):1077-87. doi: 10.1093/sleep/27.6.1077. PMID 15532201
- [Background] Hallbeck MS, Lowndes BR, Bingener J, Abdelrahman AM, Yu D, Bartley A, Park AE. The impact of intraoperative microbreaks with exercises on surgeons: A multi-center cohort study. Appl Ergon. 2017 Apr;60:334-341. doi: 10.1016/j.apergo.2016.12.006. Epub 2016 Dec 29. PMID 28166893
- [Background] Ker K, Edwards PJ, Felix LM, Blackhall K, Roberts I. Caffeine for the prevention of injuries and errors in shift workers. Cochrane Database Syst Rev. 2010 May 12;2010(5):CD008508. doi: 10.1002/14651858.CD008508. PMID 20464765
- [Background] Schweitzer PK, Randazzo AC, Stone K, Erman M, Walsh JK. Laboratory and field studies of naps and caffeine as practical countermeasures for sleep-wake problems associated with night work. Sleep. 2006 Jan;29(1):39-50. doi: 10.1093/sleep/29.1.39. PMID 16453980
- [Background] Van Dongen HP, Price NJ, Mullington JM, Szuba MP, Kapoor SC, Dinges DF. Caffeine eliminates psychomotor vigilance deficits from sleep inertia. Sleep. 2001 Nov 1;24(7):813-9. doi: 10.1093/sleep/24.7.813. PMID 11683484
- [Background] Garbarino S, Mascialino B, Penco MA, Squarcia S, De Carli F, Nobili L, Beelke M, Cuomo G, Ferrillo F. Professional shift-work drivers who adopt prophylactic naps can reduce the risk of car accidents during night work. Sleep. 2004 Nov 1;27(7):1295-302. doi: 10.1093/sleep/27.7.1295. PMID 15586782
- [Background] Tremaine R, Dorrian J, Lack L, Lovato N, Ferguson S, Zhou X, Roach G. The relationship between subjective and objective sleepiness and performance during a simulated night-shift with a nap countermeasure. Appl Ergon. 2010 Dec;42(1):52-61. doi: 10.1016/j.apergo.2010.04.005. Epub 2010 May 14. PMID 20471003
- [Background] Bonnefond A, Muzet A, Winter-Dill AS, Bailloeuil C, Bitouze F, Bonneau A. Innovative working schedule: introducing one short nap during the night shift. Ergonomics. 2001 Aug 15;44(10):937-45. doi: 10.1080/00140130110061138. PMID 11681794